CLINICAL TRIAL: NCT03771014
Title: EMPRESS: A Feasibility Study of Early Mobilisation Programmes in Critical Care
Brief Title: A Feasibility Study of Early Mobilisation Programmes in Critical Care
Acronym: EMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UHSEmpress
Record Dates: First submitted 2018-12-05; First posted 2018-12-10 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Critical Illness
Keywords: intensive care; physiotherapy; rehabilitation
MeSH Terms: conditions — Critical Illness | interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Feasibility study of two-arm pilot RCT, randomised 1:1 with blinded outcome assessments
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment at ICU discharge, hospital discharge and 3 month follow-up will be undertaken by an assessor, blinded to study group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobility (Experimental): Patients will receive standard physiotherapy regimen plus 2 x 30 minute rehabilitation sessions 5 days per week.
  Interventions: Other: Early mobility
- Standard care (No Intervention): Patients will receive standard physiotherapy regimen

INTERVENTIONS:
Other: Early mobility — This progressive mobility pathway commenced with passive cycling within 48 hours of intubation and ventilation and progressing through assisted cycling, active cycling, bed exercises, sitting, mobilising out of bed to walking
  Arms: Early mobility

SUMMARY:
The objective of this study is to determine the feasibility of delivering a very early mobility rehabilitation program in Intensive Care Units (ICU), within the context of a randomised controlled trial (RCT). This will inform the design of a future RCT investigating very early ICU rehabilitation in the UK National Health Service.

DETAILED DESCRIPTION:
Early ICU-based physical rehabilitation may benefit patients with acute severe respiratory failure by attenuating the development of severe and persistent weakness and impaired physical function seen in these patients.

Muscle wasting occurs early (within 12 hours) and progresses rapidly after ICU admission. Patients may suffer from consequent physical impairment for months or years following their discharge.

ICU based rehabilitation has the potential to improve physical function outcomes, through mitigating muscle wasting.

The investigators have successfully introduced a very early ICU mobility program in their institution, which results in increased ventilator free days and reduced length of ICU stay.

The primary aim is to investigate whether this method will work in other ICUs. EMPRESS will test the feasibility of running this intervention as an RCT. The results and a concurrent process evaluation will inform the design of a future, multi-centre randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute/unplanned medical admissions to the ICU.
* > 42 years old.
* Functionally independent prior to ICU admission (Barthel >80).
* In hospital for <5 days prior to intubation and ventilation.
* Intubated and ventilated for <72 hrs.
* Expected to remain ventilated for a further 48 hours.

Exclusion Criteria:

* In hospital for 5 days or more prior to ITU admission.
* Patients with acute brain or spinal cord injury.
* Known or suspected neurological / muscular impairment.
* Condition limiting use of cycle ergometer e.g. lower limb fracture / amputation.
* Not expected to survive >48hrs.
* Persistent therapy exemptions in first 3 days of mechanical ventilation.
* Body habitus such as unable to use cycle ergometer.
* Consultant clinician view that patient not suitable or not expected to survive admission.

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Physical Function ICU Test-scored | Up to 28 days
  This is a reliable and valid 4 item scale ( arm strength, leg strength, ability to stand and step cadence),with a score range of 0-10 and is responsive to change and predictive of key outcomes.

SECONDARY OUTCOMES:
Medical Research Council Manual Muscle Test Sum Score ( MRC-ss) | Up to 28 days
  Test of muscle strength and function, where full strength is defined as a score of 60/60 and ICU-AW as a score of <48/60
Hand held dynamometry (HHD) | Up to 12 weeks
  Assessment of hand grip strength
Chelsea Critical Care Physical Assessment tool (CPAX) | Up to 28 days
  This validated tool reliably grades physical morbidity from complete
  dependence on admission though progressive independence. Scores on ICU discharge may predict recovery trajectory.
ICU Mobility Scale | Up to 28 days
  Best level of function achieved in ICU using an 11-point ordinal scale
Timed up and go | Up to 6 months
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Clinical Frailty Score | Up to 6 months
  An 8 point score to classify patients as fit, vulnerable or frail and correlates with outcome in both elderly and younger patients. Pre illness frailty will be assessed by proxy on admission from information gathered from family member /NOK and from patient at the 3 follow-up assessment
Barthel Index for Activities of Daily Living | Up to 6 months
  Barthel ADL index is an ordinal scale used to measure performance in activities of daily living (ADL).
  Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Six minute walk test | Up to 6 months
  Widely used to assess functional exercise capacity in patients following an ICU admission
The Hospital Anxiety and Depression Scale - HADS | 6 months
  Measure of anxiety and depression in general medical population of patients. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | 6 months
  A generic assessment instrument for health and disability
EQ-5D-5L | 6 months
  The descriptive system comprises self-assessment of five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cusack, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results manuscript will be de-identified and shared on request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be addressed to EMPRESS@uhs.nhs.uk

REFERENCES:
- [Derived] Cusack R, Bates A, Mitchell K, van Willigen Z, Denehy L, Hart N, Dushianthan A, Reading I, Chorozoglou M, Sturmey G, Davey I, Grocott M. Improving physical function of patients following intensive care unit admission (EMPRESS): protocol of a randomised controlled feasibility trial. BMJ Open. 2022 Apr 15;12(4):e055285. doi: 10.1136/bmjopen-2021-055285. PMID 35428629